CLINICAL TRIAL: NCT01115894
Title: Naltrexone and CBT for Problem-Drinking MSM
Brief Title: Medication and Counseling for Controlled Drinking
Acronym: ProjectSMART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Jon Morgenstern, Ph.D., Principle Investigator, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: AA015553-01A1S1
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Alcohol Dependence; Alcohol Abuse
Keywords: problem drinking; alcohol
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- active medication + psychotherapy (Experimental)
  Interventions: Drug: Naltrexone; Behavioral: Modified Behavioral Self-Control Psychotherapy
- placebo + psychotherapy (Experimental)
  Interventions: Behavioral: Modified Behavioral Self-Control Psychotherapy; Drug: Placebo
- active medication+brief supportive counseling (Experimental)
  Interventions: Drug: Naltrexone; Behavioral: Brief Behavioral Compliance Enhancement Therapy
- placebo + brief supportive counseling (Experimental)
  Interventions: Behavioral: Brief Behavioral Compliance Enhancement Therapy; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 100 mg oral dosage daily for 12 weeks
  Arms: active medication + psychotherapy; active medication+brief supportive counseling
Behavioral: Modified Behavioral Self-Control Psychotherapy — Moderation- and cognitive-behaviorally-based psychotherapy. Treatment goal of moderation of alcohol consumption. 12 weekly, 1-hour sessions.
  Arms: active medication + psychotherapy; placebo + psychotherapy
Behavioral: Brief Behavioral Compliance Enhancement Therapy — Brief supportive counseling to enhance compliance with medication and encourage goal-setting concerning alcohol consumption.
  Arms: active medication+brief supportive counseling; placebo + brief supportive counseling
Drug: Placebo — Placebo
  Arms: placebo + brief supportive counseling; placebo + psychotherapy

SUMMARY:
Problem drinking gay and bisexual men who try to quit drinking are at risk for relapse to heavy or problematic drinking because their social lives and social outlets are often strongly associated with alcohol. These men are most receptive to interventions focused on moderation of drinking rather than abstinence. However moderation-oriented cognitive-behavior therapy (CBT) and naltrexone (NTX) are both well established treatments for problem drinkers who wish to moderate, rather than stop, drinking. Research suggests that combining these treatments may enhance their efficacy.

This study combines moderation-oriented CBT with NTX in the treatment of problem drinking gay and bisexual men, who do not wish to abstain from alcohol, to evaluate their efficacy alone and in combination. We also propose to utilize new data collection technology, Interactive Voice Response, to collect data on daily relations among drinking, sexual behavior and psychological variables thought to mediate treatment response. Our objectives are to evaluation the efficacy of 12 weeks of randomly assigned treatment, with 100 mg of NTX or placebo, combined with brief supportive therapy or modified, behavioral self-control therapy specifically tailored to gay/bisexual men; to evaluate conditional relationships between heavy drinking and likelihood of HIV risk behavior; and to evaluate daily associations among mood, craving, self-efficacy, motivation, and drinking. Assessments will include baseline, 3, 6, & 9 month follow-up. A substudy of the treatment trial will be conducted to collect and bank samples from blood for research aimed at associating naturally occurring differences in DNA with patient response to NTX, and with potential mediational mechanisms of action of NTX. Information gathered on genes or gene products may be used in conjunction with data on clinical psychological factors obtained as part of the clinical trial to evaluate relationships among genetic variants, drug effects, and mechanisms of treatment response. Patients will be asked to give a blood sample at Week 0 of the clinical trial for the purpose of carrying out genetic research.

ELIGIBILITY:
Inclusion Criteria:

* Currently sexually active with other men
* Report drinking at levels substantially in excess of established guidelines for non-hazardous drinking
* Willing to reduce drinking to non-hazardous levels
* English literate (8th grade level)

Exclusion Criteria:

* Current physical disease or condition making participant inappropriate for a medication trial, including total bilirubin elevation >110% AST or ALT elevations >300%
* History of serious psychiatric illness (psychotic disorder, bipolar disorder, or psychiatric illness requiring hospitalization)
* Recent (past three month) initiation of psychotropic medication or psychotherapy, or recent change in psychotropic medication treatment
* Current DSM-IV diagnosis of drug (other than nicotine) dependence, or lifetime diagnosis of opioid dependence
* DSM-IV alcohol dependence diagnosis judged clinically severe, history or present evidence of significant alcohol withdrawal symptoms, or recurrent use of alcohol to alleviate withdrawal
* Regular use of opioids in the past month
* History of of hypersensitivity to NTX
* Considered by study physician not to be suitable for receipt of an investigational drug
* Likely to require treatment with opiate pain medication during the course of the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Quantity of alcohol use | 9 months
Frequency of binge drinking | 9 months

SECONDARY OUTCOMES:
Frequency of HIV risk behavior | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia Addiction Services and Psychotherapy Intervention Research, New York, New York, United States